CLINICAL TRIAL: NCT05392062
Title: Pathophysiology of Gas Exchange and Time Course Changes in Spontaneously Breathing Patients With Acute Respiratory Failure Due to COVID-19. A Multicenter Prospective Study.
Acronym: COVAQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PO21075
Record Dates: First submitted 2021-08-09; First posted 2022-05-26 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Respiratory Insufficiency
Keywords: Gas exchange; COVID-19; acute respiratory distress syndrome; spontaneous breathing; Respiratory failure
MeSH Terms: conditions — Respiratory Insufficiency; COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Respiratory insufficiency (Other): Subject with respiratory insufficiency
  Interventions: Other: Pathophysiology of gas exchange

INTERVENTIONS:
Other: Pathophysiology of gas exchange — Exploration of pathophysiology of gas exchange

SUMMARY:
The pathophysiology of SARS-COV-2 related respiratory disease is still poorly understood, especially in its most severe form called acute respiratory distress syndrome (ARDS). In this case, very few studies have investigated changes in gas exchange during COVID-19 progression in spontaneously breathing patients. The investigators purpose in this study to explore the pathophysiology of gas exchange and time course changes in spontaneously breathing patients with acute respiratory failure due to COVID-19. Moreover, our aim is to identify early markers associated with worsening respiratory failure and requiring endotracheal intubation.

ELIGIBILITY:
inclusion criteria :

* Patients with a COVID-19 confirmed infection.
* Admission in intensive care unit for an acute respiratory failure requiring oxygen flow above 6l/min by facial mask.
* Presence of an arterial catheter for blood sampling.

exclusion criteria :

* Patients on mechanical ventilation on admission to the ICU.
* Patients requiring immediate intubation on admission.
* Patients admitted to the ICU for more than 48 hours at the time of inclusion.
* Pulmonary embolism diagnosed before admission to the ICU.
* Minor patients
* Pregnant women
* Patients under curatorship or guardianship
* Persons deprived of liberty by a judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2021-06-09 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
Association between measurement of intrapulmonary right-to-left shunt, ventilatory ratio and need to intubation. | Lenght of hospital stay in intensive care unit
  From date of admission in intensive care unit (ICU) until the date of death or disharge from ICU, assessed up to 90 days

SECONDARY OUTCOMES:
Association between measurement of intrapulmonary right-to-left shunt, ventilatory ratio and mortality at D90. | Day 90
  No provided
Association between measurement of intrapulmonary right-to-left shunt, ventilatory ratio and mortality at D28. | Day 28
  No provided
Association between intrapulmonary right-to-left shunt, ventilatory ratio with percentage of lung damage on chest CT-scan. | At admission
  No provided

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France